CLINICAL TRIAL: NCT06266923
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Initial Efficacy of SPH6516 Tablets in Subjects With Advanced Solid Tumors.
Brief Title: A Clinical Study of SPH6516 Tablets in the Treatment of Advanced Solid Tumors.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH6516-101
Record Dates: First submitted 2024-01-29; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPH6516 tablets (Experimental)
  Interventions: Drug: SPH6516 tablets

INTERVENTIONS:
Drug: SPH6516 tablets — SPH6516 tablets ： Orally, once daily, 25-200mg, 28 days a cycle

SUMMARY:
To evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of SPH6516 tablets in the treatment of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced solid tumors;
2. The ECOGscore is 0 to 1.
3. Expected survival ≥3 months.
4. Good organ function before first use of the investigational drug.
5. Any toxicity associated with previous antitumor therapy must have returned to ≤ grade 1.
6. Voluntarily participate in this clinical trial, understand the research procedures and be able to sign the informed consent in person.

Exclusion Criteria:

1. Subjects who have received certain treatment in the prescribed period prior to their first medication;
2. Subjects who have undergone major surgery within 6 weeks before the first medication, or who plan to undergo major surgery within 12 weeks after the first medication;
3. Subjects who have participated in any other clinical trials and received treatment within 4 weeks prior to the first medication;
4. Subjects with third space fluid accumulation that cannot be controlled by drainage or other methods; Subjects with factors affecting drug administration and absorption;
5. Subjects with allergic constitution or a history of severe allergies;
6. Subjects with active hepatitis B virus (HBV) infection, active hepatitis C virus (HCV) infection, or a history of immunodeficiency;
7. Subjects with a history or evidence of high risk cardiovascular disease;
8. Subjects with severe lung disease;
9. Pregnant and lactating female subjects; Female subjects of childbearing age or male subjectswith fertile partners who were unwilling to take effective contraceptive measures throughout the entire trial period;
10. Subjects with a clear history of neurological or psychiatric disorders;
11. Other situations in which the investigator did not consider it appropriate to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
MTD（Maximum tolerated dose） | Approximately 2 years
  Maximum tolerated dose

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Approximately 2 years
  Adverse event type, incidence, duration
Peak Plasma Concentration (Cmax） | Approximately 2 years
  PK (Pharmacokinetics)
Peak time（Tmax） | Approximately 2 years
  PK (Pharmacokinetics)
Area under the plasma concentration versus time curve (AUC) | Approximately 2 years
  PK (Pharmacokinetics)
half-life（T1/2） | Approximately 2 years
  PK (Pharmacokinetics)
Objective response rate(ORR) | Approximately 2 years
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1
Progression-free survival (PFS) | Approximately 2 years
  The interval between the date of the first dose of trial treatment until first documentation of disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Ruijin Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai